CLINICAL TRIAL: NCT04729387
Title: EPIK-O: A Phase III, Multi-center, Randomized (1:1), Open-label, Active-controlled, Study to Assess the Efficacy and Safety of Alpelisib (BYL719) in Combination With Olaparib as Compared to Single Agent Cytotoxic Chemotherapy, in Participants With no Germline BRCA Mutation Detected, Platinum-resistant or Refractory, High-grade Serous Ovarian Cancer
Brief Title: Alpelisib Plus Olaparib in Platinum-resistant/Refractory, High-grade Serous Ovarian Cancer, With no Germline BRCA Mutation Detected
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719K12301; 2024-510782-42-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: Alpelisib; olaparib; paclitaxel; pegylated liposomal doxorubicin; high grade; serous ovarian; fallopian or peritoneal cancer; no germline BRCA mutation; BRCA wild type; platinum-resistant or refractory; prior PARP inhibitor exposure; EPIK-O
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Alpelisib; olaparib; Paclitaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alpelisib+olaparib (Experimental): Alpelisib 200 mg orally once daily and olaparib 200 mg orally twice daily on a continuous dosing schedule.
  Interventions: Drug: Alpelisib; Drug: Olaparib
- Paclitaxel or PLD (Active Comparator): Investigator's choice of one of 2 single agent cytotoxic chemotherapies: Paclitaxel 80 mg/m2 intravenously weekly or Pegylated liposomal Doxorubicin (PLD) 40-50 mg/m2 (physician discretion) intravenously every 28 days.
  Interventions: Drug: Paclitaxel; Drug: Pegylated liposomal doxorubicin (PLD)

INTERVENTIONS:
Drug: Alpelisib — Alpelisib will be administered at 200 mg orally once daily following food on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28-day cycle
  Other Names: BYL719
  Arms: Alpelisib+olaparib
Drug: Olaparib — Olaparib will be administered at 200 mg orally twice daily irrespective of meals on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28-day cycle.
  Arms: Alpelisib+olaparib
Drug: Paclitaxel — Paclitaxel will be administered at 80 mg/m2 as an intravenous infusion weekly during a 28-day treatment cycle, starting on Cycle 1 Day 1, and on Day 8, Day 15 and Day 22 of every cycle thereafter
  Arms: Paclitaxel or PLD
Drug: Pegylated liposomal doxorubicin (PLD) — PLD will be administered at 40-50 mg/m2 (physician discretion) as an intravenous infusion once every 28-days in a 28 day treatment cycle, starting on Cycle 1 Day 1
  Arms: Paclitaxel or PLD

SUMMARY:
The objective of this study is to assess the efficacy and safety of the combination of alpelisib and olaparib compared with single agent cytotoxic chemotherapy in patients with platinum resistant or refractory high-grade serous ovarian cancer, with no germline BRCA mutation detected.

DETAILED DESCRIPTION:
This study will include adult women with platinum resistant or refractory high-grade serous ovarian cancer, with no germline BRCA mutation detected. Participants will be randomized in a 1:1 ratio to either alpelisib plus olaparib or single agent cytotoxic chemotherapy (paclitaxel or PLD) in this open-label, active controlled study.

Participants will continue to receive study treatment until disease progression, unacceptable toxicity that precludes further treatment, or until discontinuation of study treatment due to any other reason. After treatment discontinuation, all participants will enter in the post-treatment follow-up period, which consists of a safety follow-up visit and a 9-week post-progression visit. Once they complete the post-treatment follow-up, participants will then enter the survival follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has histologically confirmed diagnosis of high-grade serous or high-grade endometrioid ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
* Measurable disease, i.e., at least one measurable lesion per RECIST 1.1 criteria (a lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation)
* If no measurable disease is present, the disease should be assessable by Gynecologic Cancer Intergroup criteria (GCIC) for CA-125
* Participant has no germline BRCA1/2 mutation as determined by an FDA-approved assay
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participant has platinum-resistant (progression within one to six months after completing platinum-based therapy) or platinum refractory disease (progression during treatment or within 4 weeks after the last dose), where platinum-based therapy is not an option, according to the GCIG 5th Ovarian Cancer Consensus Conference definitions (Wilson et al 2016). The platinum-based chemotherapy regimen does not necessarily need to be the last regimen the participant received prior to study entry
* Participant must have received at least one but no more than three prior systemic treatment regimens and for whom single-agent chemotherapy is appropriate as the next line of treatment
* Participant has received prior bevacizumab or is not eligible to receive bevacizumab due to medical reasons.

Key Exclusion Criteria:

* Participant has received prior treatment with any PI3K, mTOR or AKT inhibitor
* Participant is concurrently using other anti-cancer therapy
* Participant is in a state of small or large bowel obstruction or has other impairment of gastrointestinal (GI) function or GI disease
* Participant has had surgery within 14 days prior to starting study drug or has not recovered from major adverse effects
* Participant has not recovered from all toxicities related to prior anticancer therapies to baseline or NCI CTCAE Version 4.03 Grade ≤1. Exception to this criterion: participants with any grade of alopecia are allowed to enter the study
* Participant has an established diagnosis of diabetes mellitus type I or uncontrolled type II based on fasting plasma glucose and HbA1c
* Participants with liver impairment and Child Pugh score B or C
* Participant has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to randomization, and who has not recovered to baseline, grade 1 or better from related adverse effects of such therapy (with the exception of alopecia)
* Participant has a known hypersensitivity to any of the study drugs or excipients
* Participant has a history of myelodysplastic syndrome or acute myeloid leukemia, or presents clinical and/ or laboratory features suggestive thereof.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women
Enrollment: 358 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) based on Blinded Independent Review Committee (BIRC) assessment using RECIST 1.1 criteria | From randomization until the date of the first documented progression or death due to any cause, whichever comes first, assessed up to approximately 23 months
  Progression-free survival (PFS) was defined as the time from randomization until the first documented disease progression or death from any cause, based on BIRC assessment. Participants without an event were censored at the date of their last adequate tumor assessment. Clinical deterioration without objective radiologic evidence was not considered disease progression in the primary efficacy analysis.

SECONDARY OUTCOMES:
Overall survival | From randomization until death, assessed up to approximately 44 months
  Overall survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive
Overall Response Rate (ORR) with confirmed response based on BIRC assessment according to RECIST 1.1 criteria | Up to approximately 23 months
  Overall response rate (ORR) with confirmed response was defined as the percentage of participants whose best overall response (BOR) was a confirmed complete response (CR) or confirmed partial response (PR), as determined by BIRC according to RECIST 1.1 criteria.
Clinical benefit rate (CBR) with confirmed response based on BIRC assessment according to RECIST 1.1 | Up to approximately 23 months
  Clinical benefit rate (CBR) with confirmed response was defined as the percentage of participants whose best overall response was a confirmed CR or PR, or stable disease (SD) maintained for at least 24 weeks. CR, PR, and SD were determined by BIRC according to RECIST 1.1 criteria.
Time to response (TTR) based on BIRC assessment and according to RECIST 1.1 | From the date of randomization to the first documented response, assessed through Month 12
  Time to response (TTR) was defined as the interval from randomization to the first documented occurrence of either complete response (CR) or partial response (PR), which was subsequently confirmed (using the date of initial response, not the confirmation date). CR and PR were determined based on tumor response data assessed by BIRC according to RECIST 1.1 criteria.
Duration of response (DOR) with confirmed response based on BIRC assessment and according to RECIST 1.1 | From first documented response to first documented progression or death, assessed up to approximately 23 months
  Duration of response (DOR) with confirmed response was calculated only for participants whose best overall response was a confirmed complete response (CR) or confirmed partial response (PR), based on tumor response data assessed by BIRC according to RECIST 1.1. The start date was the date of the first documented CR or PR (i.e., the initial response date, not the confirmation date), and the end date was the date of first documented disease progression or death due to underlying cancer. Participants without progression or cancer-related death were censored at the date of their last adequate tumor assessment.
Time to definitive deterioration of the Eastern Cooperative Oncology Group (ECOG) performance status (PS) | Up to approximately 18 months
  Performance status (PS) was evaluated using the ECOG scale, which comprises six grades (0 to 5), where 0 represents fully active and 5 represents death. Time to definitive deterioration in ECOG PS was defined as the interval from randomization to the date when ECOG PS worsened by at least one category from baseline and remained worsened. Deterioration was considered definitive if there was no subsequent improvement to the baseline category or better. Participants were censored if no definitive deterioration occurred before the earlier of: (i) the analysis cut-off date or (ii) initiation of a new anti-neoplastic therapy. The censoring date was the date of the last PS assessment prior to the cut-off or start of new therapy.
Number of participants with dose interruptions and dose reductions | From randomization until end of treatment, assessed up to approximately 18 months
  The number of participants with dose reductions/interruptions was assessed and summarized by study treatment.
Dose intensity | From randomization until end of treatment, assessed up to approximately 18 months
  Dose intensity was computed as the ratio of actual cumulative dose received to actual duration of exposure and summarized by study treatment.
Area under the curve calculated to the end of a dosing interval (tau) at steady-state (AUCtau) of alpelisib and olaparib | Day 8 Cycle 1 (pre-dose, 1, 2, 3, 4, 6, 8 and 24 hours post dose), Day 1 on Cycle 2, 4 and 8 (pre-dose)
  The AUCtau will be assessed to characterize the pharmacokinetics of alpelisib when administered in combination of olaparib
Area under the curve from time zero to the last measurable concentration sampling time (AUClast)of alpelisib and olaparib | Day 8 Cycle 1 (pre-dose, 1, 2, 3, 4, 6, 8 and 24 hours post dose), Day 1 on Cycle 2, 4 and 8 (pre-dose)
  The AUClast will be assessed to characterize the pharmacokinetics of alpelisib when administered in combination of olaparib
Maximum Concentration (Cmax) of alpelisib and olaparib | Day 8 Cycle 1 (pre-dose, 1, 2, 3, 4, 6, 8 and 24 hours post dose), Day 1 on Cycle 2, 4 and 8 (pre-dose)
  The Cmax will be assessed to characterize the pharmacokinetics of alpelisib when administered in combination of olaparib
Time to reach maximum concentration (Tmax) of alpelisib and olaparib | Day 8 Cycle 1 (pre-dose, 1, 2, 3, 4, 6, 8 and 24 hours post dose), Day 1 on Cycle 2, 4 and 8 (pre-dose)
  The Tmax will be assessed to characterize the pharmacokinetics of alpelisib when administered in combination of olaparib
Change from baseline in Function Assessment of Cancer Therapy-Ovarian Trial Outcome Index (FACT-O TOI) | Baseline, then every 8 weeks for 18 months, every 12 weeks thereafter until RECIST 1.1 progression, death, consent withdrawal, loss to follow-up, participant/guardian decision, and at End of Treatment (EOT) within 14 days from last dose.
  The Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) combines scores from Physical Well-Being (PWB), Functional Well-Being (FWB), and the Ovarian Cancer Subscale (OCS). Each item is rated on a 0-4 Likert scale (0 = 'Not at all', 4 = 'Very much'). The TOI score is the sum of these subscales and ranges from 0 to 100, with higher scores reflecting better quality of life and physical/functional status. A positive change from baseline indicates improvement in physical/functional well-being and ovarian cancer-specific symptoms, while a negative change indicates deterioration in these domains.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (89):
- United States (16):
  - Arizona Oncology Associates, Phoenix, Arizona
  - HonorHealth, Phoenix, Arizona
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Maryland Oncology Hematology P A, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - University Of Cincinnati, Cincinnati, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology P A, Bedford, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology P A, San Antonio, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Caba
- Australia (3):
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Shepparton, Victoria
  - Novartis Investigative Site, Sydney
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Namur
- Brazil (2):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (4):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- China (5):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense C
- Finland (3):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (5):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
- Italy (6):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Napoli
- Malaysia (4):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (2):
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mexico City
- Novartis Investigative Site, Eindhoven, Netherlands
- Portugal (2):
  - Novartis Investigative Site, Loures
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Arkhangelsk, Russia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Bratislava, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Izmir, Karsiyaka
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Adana, Yuregir
  - Novartis Investigative Site, Ankara
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Konstantinopoulos PA, Gonzalez-Martin A, Cruz FM, Friedlander M, Glasspool R, Lorusso D, Marth C, Monk BJ, Kim JW, Hinson P, Ajipa O, Pretre V, Han Y, Matulonis UA. EPIK-O/ENGOT-OV61: alpelisib plus olaparib vs cytotoxic chemotherapy in high-grade serous ovarian cancer (phase III study). Future Oncol. 2022 Oct;18(31):3481-3492. doi: 10.2217/fon-2022-0666. Epub 2022 Sep 6. PMID 36066851